CLINICAL TRIAL: NCT06470269
Title: Examining Clinical Reasoning With Eye Tracking
Brief Title: Examining Clinical Reasoning With Eye-tracking
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00102074
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Diagnosis; Educational Problems
Keywords: Eye tracking; Clinical Reasoning; Cognitive Development
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Expert: Physicians
  Interventions: Behavioral: Eye tracking
- Novice: Medical Students
  Interventions: Behavioral: Eye tracking

INTERVENTIONS:
Behavioral: Eye tracking — Recording the eye movement of participants while they read medical cases.

SUMMARY:
The process of medical information intake, interpretation and diagnosis, commonly referred to as clinical reasoning, involves a complex interaction between visual perception and multiple cognitive processes. Assessing students' clinical reasoning skills is a challenging but critical task in developing an optimal teaching curriculum. In this project, the investigators plan to apply the eye-tracking technology to medical education with a specific goal of examining cognitive processing during reading medical chart and x-ray films. Data collected by eye tracking technology will help investigate the perceptual and cognitive underpinnings of clinical reasoning (CR), misinterpretation and misdiagnosis among three participant groups with different levels of clinical experience. Knowledge gained from this project will help to decode the intricate cognitive loop involved in medical interpretation. Further, this study will help to develop alternative methods of assessing student's clinical reasoning skills and promote medical education with novel eye tracking technology.

DETAILED DESCRIPTION:
Objective:

In this project, the investigators plan to apply the eye-tracking technology to medical education with a specific goal of examining cognitive processing during clinical reasoning (CR). The investigators expect that by checking the eye movements of medical trainees during case and image reading, a list of valid behavioral markers could be created, to quantitatively classify the expertise, identify the moment of decision-making difficulty, and decode the source of the judgement errors. To examine differences in CR processes across varying levels of expertise, three categories of participants (novice, intermediate, and expert) will be recruited. While participants' eye motions are tracked, participants will read a trauma case, provide a diagnosis and propose a suitable treatment plan. The investigators postulate that 1) different participant groups will produce significantly different CR outcomes, measured by their score on diagnostic judgement and treatment plan; 2) participants will display different gaze fixation patterns; and 3) combining evidence from clinical judgement and eye behavior analysis will provide useful information regarding the source of judgment errors.

Research Method/Procedures:

Staff and students in the SSRL (Surgical Simulation Research Lab) with a difficulty level of health training background will be enrolled as participants in the study. A trauma case with complex life-threatening situations will be presented. The case is a trauma cases with multiple internal injuries. The case will be summarized into a one-page description and 3 x-ray films. Our participants will need to make a diagnosis and give a treatment plan based on case information displayed on a screen. The total reading time will be 4 minutes. During the case reading, the Tobii X2-60, a high-resolution remote eye-tracker, will be used to capture the participant's eye movements. In addition, the investigators will develop a 15-20 quiz regarding the patient's condition and the participant's final diagnosis. The total score and errors in the quiz will be used to describe participants' overall quality of their clinical reasoning.

The investigators will carefully examine participants' eye motions and report their scanning patterns during case reading. Specifically, the investigators will look for moments when participants rapidly move their eyes (saccade) over a sentence before fixating on a particular word (fixation). These eye behavior parameters have previous associations with mental workload and reasoning processing methods, which can be used to further analyze results.

Plan for Data Analysis:

The investigators will firstly compare quiz scores and eye behaviors variables across the three participant groups with different clinical experience levels. The investigators will then analyze eye-scanning patterns on case readings across the three different groups. Specifically, The investigators predict that experts will achieve the highest score in quiz. The investigators therefore will examine the expert's short and long fixation locations over the case reading. The assumption is that experts know where to find key information in the case description and mentally connect separate information together to generate an correct judgement in the short period of time. Fixation spots recorded from the novice and intermediate groups will be compared with experts'. Differences will help us identify different visual searching strategies over different stages in the development of clinical reasoning skills. Lastly, the investigators will examine clinical judgement errors and check the root cause by connecting quiz errors with eye behaviors. If a participant failed to give a long fixation to key case features in the case description, the clinical decision error may be due to a checking problem. If a participant performs a long fixation to key case features, the clinical decision error may due to recognition or decision-making problems.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Has normal or corrected to normal vision
* Healthcare provider

Exclusion Criteria:

-Non healthcare provider

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physicians in neurology department and medical students registered in medical school.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Eye Fixation | During case reading (about 5 minutes)
  Eye fixation over key reading area

SECONDARY OUTCOMES:
Eye Saccade | During case reading (about 5 minutes)
  Rapid eye shift between key reading areas

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No